CLINICAL TRIAL: NCT02187744
Title: A RANDOMIZED, DOUBLE-BLIND PHARMACOKINETIC STUDY OF PF-05280014 PLUS TAXOTERE (REGISTERED) AND CARBOPLATIN VERSUS HERCEPTIN (REGISTERED) PLUS TAXOTERE (REGISTERED) AND CARBOPLATIN FOR THE NEOADJUVANT TREATMENT OF PATIENTS WITH OPERABLE HER2-POSITIVE BREAST CANCER
Brief Title: A Study Of PF-05280014 Or Trastuzumab Plus Taxotere® And Carboplatin In HER2 Positive Breast Cancer In The Neoadjuvant Setting (REFLECTIONS B327-04)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3271004; REFLECTIONS B327-04; 2013-004679-11 (EudraCT Number); REFLECTIONS (B327-04) (Other: Alias Study Number)
Record Dates: First submitted 2014-06-30; First posted 2014-07-11 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Early Breast Cancer
Keywords: Biosimilars; Non-inferiority; Neoadjuvant Setting; Early Breast Cancer; PK; Phase 3; Trastuzumab; Herceptin; HER2 Positive
MeSH Terms: conditions — Breast Neoplasms | interventions — PF-05280014; Docetaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-05280014 (Experimental)
  Interventions: Biological: PF-05280014; Drug: Taxotere®; Drug: Paraplatin®
- Herceptin® (Active Comparator)
  Interventions: Biological: Trastuzumab-EU; Drug: Taxotere®; Drug: Paraplatin®

INTERVENTIONS:
Biological: PF-05280014 — Concentrate for solution for infusion, sterile vial 150 mg, Day 1 Cycle 1 will be a loading dose of 8 mg/kg infused over 90 minutes. Subsequent infusions will follow every 3 weeks (i.e., cycled every 21 days) with a dose of 6 mg/kg administered over 30 to 90 minutes depending on tolerability, maximum of 6 cycles.
  Arms: PF-05280014
Drug: Taxotere® — Injection concentrate single-dose vials containing 20 mg (0.5 mL) or 80 mg (2 mL), each mL contains 40 mg docetaxel (anhydrous) and 1040 mg polysorbate 80, The starting dose of Taxotere® (docetaxel) will be 75 mg/m2 administered intravenously over 60 minutes every three weeks on Day 1 of each cycle (i.e., every 21 days), maximum 6 cycles.
  Other Names: docetaxel
  Arms: PF-05280014
Drug: Paraplatin® — Lyophilized powder, single-dose vials containing 50 mg, 150 mg, and 450 mg of Carboplatin for administration by intravenous infusion (each vial contains equal parts by weight of Carboplatin and mannitol), starting dose 6 AUC, over 15 minutes or longer every three weeks on Day 1 of each cycle (i.e., every 21 days), maximum 6 cycles.
  Other Names: carboplatin
  Arms: PF-05280014
Biological: Trastuzumab-EU — Concentrate for solution for infusion, sterile vial 150 mg, Day 1 Cycle 1 will be a loading dose of 8 mg/kg infused over 90 minutes. Subsequent infusions will follow every 3 weeks (i.e., cycled every 21 days) with a dose of 6 mg/kg administered over 30 to 90 minutes depending on tolerability, maximum 6 cycles.
  Arms: Herceptin®
Drug: Taxotere® — Injection concentrate single-dose vials containing 20 mg (0.5 mL) or 80 mg (2 mL), each mL contains 40 mg docetaxel (anhydrous) and 1040 mg polysorbate 80, The starting dose of Taxotere® (docetaxel) will be 75 mg/m2 administered intravenously over 60 minutes every three weeks on Day 1 of each cycle (i.e., every 21 days), maximum 6 cycles.
  Other Names: docetaxel
  Arms: Herceptin®
Drug: Paraplatin® — Lyophilized powder, single-dose vials containing 50 mg, 150 mg, and 450 mg of Carboplatin for administration by intravenous infusion (each vial contains equal parts by weight of Carboplatin and mannitol), starting dose 6 AUC, over 15 minutes or longer every three weeks on Day 1 of each cycle (i.e., every 21 days), maximum 6 cycles.
  Other Names: carboplatin
  Arms: Herceptin®

SUMMARY:
The current study will compare PK, efficacy, safety, and immunogenicity of PF-05280014 (Trastuzumab-Pfizer) in combination with Taxotere® and Carboplatin (Paraplatin) versus Herceptin® (Trastuzumab-EU) approved in the EU in combination with Taxotere® and Carboplatin (Paraplatin) in patients with operable HER2 positive, breast cancer in the neoadjuvant setting. The hypothesis to be tested in this study is the percentage of patients with steady state Cycle 5 Ctrough (Cycle 6 pre-dose) >20 µg/mL of trastuzumab-Pfizer is similar to EU-approved trastuzumab, using a margin of -12.5%.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2 overexpressing invasive breast cancer.
* Plan for definitive surgical resection of breast tumor (i.e., lumpectomy or mastectomy, and sentinel node (SN) biopsy or axillary lymph node dissection (ALND).
* Plan for neoadjuvant chemotherapy.
* Measurable disease in the breast after diagnostic biopsy, defined as longest diameter ≥ 2.0 cm.

Exclusion Criteria:

* Bilateral breast cancer.
* Inflammatory breast cancer.
* Presence of known distant metastases.
* Received prior treatment, including chemotherapy, endocrine therapy, biologic therapy, radiation or surgery with the exception of diagnostic biopsy for primary breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 226 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2016-03-09 (Actual); Study Completion 2016-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (4):
  - Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Millennium Oncology (Imaging Facility), Kingwood, Texas
  - Millennium Oncology (Imaging Facility), Shenandoah, Texas
  - Millennium Oncology, Shenandoah, Texas
- SI 'Republican Research and Practice Centre of Oncology and Medical Radiology n.a. N.N. Alexandrov', Lyasny, Minsk Oblast, Belarus
- Fakultni nemocnice Hradec Kralove, Hradec Králové, Czechia
- Hungary (6):
  - Bacs-Kiskun Megyei Korhaz, Kecskemét, Bács-Kiskun county
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar-I. sz. Belgyogyaszati Klinika Onkologiai Reszleg, Budapest
  - Szent Imre Egyetemi Oktato Korhaz, Budapest
  - Uzsoki Utcai Korhaz, Onkoradiologia, Sugarterapia Fovarosi Onkoradiologiai Kozpont, Budapest
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktatokorhaz,, Miskolc
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz - Rendelointezet, Szolnok
- Italy (4):
  - Division of Medical Senology, Milan, MI
  - Divisione di Oncologia Medica B, Roma, RM
  - IRCCS Istituto Nazionale Tumori Regina Elena (IRE), Roma, RM
  - Dept. of Surgery, Roma, RM
- Poland (3):
  - Szpitale Wojewodzkie w Gdyni Sp. z o.o., Oddzial Onkoligii i Radioterapii, Gdynia
  - Oddzial Chorob Rozrostowych, Lodz
  - SPZOZ MSW z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
- Russia (19):
  - State Budgetary Healthcare Institution "Leningrad Regional Oncological Dispensary", Kuzmolovo, Leningradskaya Oblast'
  - "State Budgetary Healthcare Institution ""Republican Clinical Oncological Dispensary of the Ministry, Ufa, Republic Bashkortost
  - Regional Budgetary Healthcare Institution "Kursk regional clinical oncological Dispensary", Kislino Settlement, Ryshkovskiy Village Council
  - "State Budgetary Healthcare Institution of Stavropol Region ""Pyatigorsk Oncological Dispensary""", Pyatigorsk, Stavropol Kray
  - State Budgetary Healthcare Institution "Volgograd Regional Oncological Dispensary #3", Volzhsky, Volgograd Oblast
  - SBHI "Regional Oncology Dispensary", Irkutsk
  - Regional Budgetary Healthcare Institution, Kursk
  - FSBI "Russian Oncology Scientific center n.a. N. N. Blokhin" RAMS, Moscow
  - State Budgetary Institution Of Healthcare, Moscow
  - SBHI of NNR "Clinical diagnostic center", Nizhny Novgorod
  - State Budgetary Healthcare Institution of NNR "Nizhniy Novgorod Regional Oncological Dispensary", Nizhny Novgorod
  - Budgetary Institution of healthcare of Omsk region "Clinical oncological dispensary", Omsk
  - State Budgetary Educational Institution of Higher Professional Education "North-Western State, Saint Petersburg
  - Saint-Peterbsurg Clinical Oncological dispensary of Moscow district, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "Oncological Dispensary of Moscow District", Saint Petersburg
  - LLC RAMSAY Diagnostic RUS, Saint Petersburg
  - "Federal State Institution ""Scientific Research Institute of Oncology n.a. N.N.Petrov"", Saint Petersburg
  - Saint-Petersburg State Budgetary Institution of healthcare "City Clinical Oncological Dispensary", Saint Petersburg
  - SRBHI "Regional Clinical Oncology Dispensary", Veliky Novgorod
- Institute For Oncology And Radiology Of Serbia, Belgrade, Serbia
- Slovakia (3):
  - Onkologicky ustav sv. Alzbety, s.r.o., Bratislava
  - Narodny Onkologicky ustav, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
- Ukraine (10):
  - Municipal Healthcare Institution 'Chernihiv Regional Oncology Dispensary', Mamology Department, Chernihiv
  - MI 'City Dnipropetrovsk Multi-field Clin. Hospital #4 of DRC', Dep.-nt of Chemotherapy;, Dnipropetrovsk
  - SI "Institute of Medical Radiology n.a.S.P. Hrygoriev of National Academy, Kharkiv
  - Munincipal Healthcare Institution"Kharkiv Regional Clinical Oncologic Center, Kharkiv
  - Khmelnytskyi Regional Oncologic Dispensary, Khmelnytskyi
  - MI 'Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional Council', Kryvyi Rih
  - Lviv State Oncologic Regional Treatment and Diagnostic Center, Lviv
  - Municipal Institution 'Odesa Regional Clinical Hospital', Mamology Center, Odesa
  - Regional Municipal Institution "Sumy Regional Clinical Oncology Dispensary", Thoracic Department, Sumy
  - Vinnytsia Regional Oncology Clinical Dispensary, Chemotherapy Department, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Lammers PE, Dank M, Masetti R, Abbas R, Hilton F, Coppola J, Jacobs I. Neoadjuvant PF-05280014 (a potential trastuzumab biosimilar) versus trastuzumab for operable HER2+ breast cancer. Br J Cancer. 2018 Aug;119(3):266-273. doi: 10.1038/s41416-018-0147-1. Epub 2018 Jul 13. PMID 30002437
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3271004&StudyName=A%20Randomized%2C%20Double-blind%20Pharmacokinetic%20Study%20Of%20Pf-05280014%20Plus%20Taxotere%20%28registered%29%20And%20Carboplatin%20Versus%20Herceptin%20%28registered%29%20Plus%20Taxotere%20%28registered%29%20And%20Carboplatin%20For%20The%20Neoadjuvant%20Treatment%20Of%20Patients%20With%20Operable%20Her2-positive%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A single participant was randomized but not treated; this participant was included in the ITT population, but not in the Participant Flow, Per Protocol, or Safety populations.
Groups:
- PF-05280014: Participants received a loading dose of 8 mg/kg of PF-05280014 on Cycle 1 Day 1. Subsequent infusions followed every 3 weeks with a dose of 6 mg/kg. Taxotere 75 mg/m2 and carboplatin area under the concentration versus time curve (AUC) 6 were administered on Day 1 of each cycle.
- Trastuzumab-EU: Participants received a loading dose of 8 mg/kg of trastuzumab-EU on Cycle 1 Day 1. Subsequent infusions followed every 3 weeks with a dose of 6 mg/kg. Taxotere 75 mg/m2 and carboplatin AUC 6 were administered on Day 1 of each cycle.
Period: Study
Arm/Group | PF-05280014 | Trastuzumab-EU
Started | 113 (Received treatment) | 112 (Received treatment)
Completed | 109 | 106
Not Completed | 4 | 6
Not completed — Participant refused further follow-up | 1 | 0
Not completed — Other | 2 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Related adverse event, not serious | 0 | 2
Not completed — Death | 1 | 0
Not completed — Related adverse event, serious non-fatal | 0 | 1
Period: Treatment
Arm/Group | PF-05280014 | Trastuzumab-EU
Started | 113 | 112
Completed | 109 | 107
Not Completed | 4 | 5
Not completed — Death | 1 | 0
Not completed — Related adverse event, serious non-fatal | 0 | 1
Not completed — Related adverse event, not serious | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 2 | 0
Not completed — Participant refused continued treatment | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized into the study.
Groups:
- PF-05280014: Participants received a loading dose of 8 mg/kg of PF-05280014 on Cycle 1 Day 1. Subsequent infusions followed every 3 weeks with a dose of 6 mg/kg. Taxotere 75 mg/m2 and carboplatin AUC 6 were administered on Day 1 of each cycle.
- Total: Total of all reporting groups
Arm/Group | PF-05280014 | Trastuzumab-EU | Total
Number analyzed (Participants) | 114 | 112 | 226
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (11.9) | 51.2 (12.7) | 52.6 (12.3)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 114 | 112 | 226

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Steady State Drug Concentration Ctrough (Cycle 6 Pre-dose) >20 µg/mL at Cycle 5.
Description: The percentage of participants with Cycle 5 Ctrough (Cycle 6 pre-dose) >20 μg/mL in each treatment group, the denominator being the number of participants in the per protocol population for each treatment group.
Time Frame: Cycle 5
Population: All participants who were HER2+ and randomized into the study; and who had received 6 cycles of PF-05280014 or trastuzumab-EU treatment; and had no temporary delays of PF-05280014 or trastuzumab-EU treatment lasting more than 1 week; and had no other significant protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 101 | 89
Percentage of participants | 92.1 [85.0 to 96.5] | 93.3 [85.9 to 97.5]
Statistical Analysis 1: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Non-Inferiority or Equivalence — The hypothesis to be tested in this study is the percentage of participants with steady state (Cycle 5) Ctrough >20 μg/mL of PF-05280014 is non-inferior to trastuzumab-EU using a margin of -12.5%; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-8.02 to 6.49], Standard Error of Mean 3.70 — Stratified analysis was based on the normal approximation to the binomial distribution, adjusting for the randomization strata of primary tumor size, estrogen receptor status and by progesterone receptor status
Statistical Analysis 2: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-8.59 to 6.23], Standard Error of Mean 3.78 — Unstratified analysis

2. Secondary Outcome: Mean Predose Trastuzumab-Pfizer and Trastuzumab-EU Concentrations at Cycles 1 Through 6.
Description: Samples of blood were taken pre-dose on Cycles 1, 2, 4, 5, and 6, and at 1 hour post dose on Cycles 1 and 5 for pharmacokinetic evaluation.
Time Frame: Cycles 1 through 6
Population: All participants who were HER2+ and randomized into the study; and who have received 6 cycles of PF-05280014 or trastuzumab-EU treatment; and had no temporary delays of PF-05280014 or trastuzumab-EU treatment lasting more than 1 week; and had no other significant protocol deviations.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 101 | 89
μg/mL
  Cycle 1/Day 1 0 hours N= 101, 88 | 2.313 (17.949) | 1.318 (12.366)
  Cycle 1/Day 1 1 hour N= 97, 80 | 160.4 (57.329) | 164.8 (47.033)
  Cycle 2/Day 21 0 hours N= 99, 88 | 24.29 (13.796) | 27.20 (10.650)
  Cycle 4/Day 63 0 hours N= 98, 89 | 33.43 (14.488) | 37.33 (15.629)
  Cycle 5/Day 84 0 hours N= 101, 87 | 35.01 (15.571) | 40.44 (26.765)
  Cycle 5/Day 84 1 hour N= 90, 80 | 137.0 (37.748) | 138.8 (37.417)
  Cycle 6/Day 105 0 hours N= 101, 89 | 37.77 (17.523) | 40.10 (16.670)

3. Secondary Outcome: Pathologic Complete Response (pCR) Defined as the Absence of Invasive Neoplastic Cells in the Breast and Lymph Nodes.
Description: Following surgery after treatment completion, tumors were assessed as Complete Pathological Response, Partial Pathological Response, or No Pathological Response.
Time Frame: Cycle 6/End of treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 100 | 86
Percentage of participants | 47.0 [36.9 to 57.2] | 50.0 [39.0 to 61.0]
Statistical Analysis 1: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Superiority or Other; Mean Difference (Final Values) = -2.81, 95% CI 2-sided [-16.58 to 10.96], Standard Error of Mean 7.03 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Superiority or Other; Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-17.40 to 11.40], Standard Error of Mean 7.35 — Unstratified analysis

4. Secondary Outcome: Objective Response Rate (ORR) Defined as the Percentage of Participants Having Complete or Partial Response at End of Treatment, Based on Radiographic Assessments of the Tumor.
Description: ORR was defined as Complete Response (CR), Partial Response (PR), Stable (SD), Progressive Disease (PD) or Indeterminate (IND). ORR was the percentage of participants who had CR or PR at Cycle 6/End of treatment.
Time Frame: Cycle 6/End of treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 101 | 89
Percentage of participants | 88.1 [80.2 to 93.7] | 82.0 [72.5 to 89.4]
Statistical Analysis 1: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Superiority or Other; Mean Difference (Final Values) = 5.96, 95% CI 2-sided [-4.01 to 15.94], Standard Error of Mean 5.09 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Superiority or Other; Mean Difference (Final Values) = 6.10, 95% CI 2-sided [-4.08 to 16.27], Standard Error of Mean 5.19 — Unstratified analysis

5. Secondary Outcome: Incidence of Anti-trastuzumab Antibodies (ADAs) at Cycles 1 Through 6.
Description: The number of participants with positive (titer >=1.00) pre-dose ADA samples, participants counted towards the total if for at least one sample, the ADA was positive.
Time Frame: Cycles 1 through 6
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Number of participants
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 113 | 112
Number of participants
  Cycle 1 (n=113,112) | 0 | 1
  Cycle 2 (n=111,112) | 0 | 0
  Cycle 4 (n=108,109) | 0 | 0
  Cycle 6 (n=108,108) | 0 | 0

6. Secondary Outcome: Incidence of Neutralizing Antibodies (NAb) at Cycles 1 Through 6.
Description: The number of participants with positive (NAb response >=1.48) pre-dose NAb samples, participants counted towards the total if for at least one sample, the NAb was positive.
Time Frame: Cycles 1 through 6
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Number of participants
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 113 | 112
Number of participants
  Cycle 1 (n=113,112) | 0 | 0
  Cycle 2 (n=110,112) | 0 | 0
  Cycle 4 (n=108,110) | 0 | 0
  Cycle 6 (n=108,108) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were captured from the beginning of the study drug treatment up to 6 months after the last dose. Treatment emergent adverse events were captured from the beginning of the study drug treatment up to 50 days after the last dose.
Description: Treatment emergent adverse events were defined as any adverse event that occurred or any preexisting adverse event that worsened within the reporting time frame.
Arm/Group | PF-05280014 | Trastuzumab-EU
Serious Adverse Events (participants affected / at risk) | 7/113 | 6/112
Other Adverse Events (participants affected / at risk) | 106/113 | 106/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05280014 (N=113) | Trastuzumab-EU (N=112)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Injection site abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05280014 (N=113) | Trastuzumab-EU (N=112)
Anaemia (Blood and lymphatic system disorders) | 56 | 51
Neutropenia (Blood and lymphatic system disorders) | 37 | 41
Leukopenia (Blood and lymphatic system disorders) | 16 | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 38 | 34
Diarrhoea (Gastrointestinal disorders) | 16 | 19
Vomiting (Gastrointestinal disorders) | 7 | 10
Asthenia (General disorders) | 36 | 23
Fatigue (General disorders) | 15 | 19
Pyrexia (General disorders) | 6 | 5
Alanine aminotransferase increased (Investigations) | 7 | 10
Aspartate aminotransferase increased (Investigations) | 3 | 7
Decreased appetite (Metabolism and nutrition disorders) | 13 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 4
Dysgeusia (Nervous system disorders) | 4 | 6
Neuropathy peripheral (Nervous system disorders) | 6 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 72 | 69

LIMITATIONS AND CAVEATS:
It was decided that the secondary study objective to explore the relationship between drug exposure and pCR for PF-05280014 versus trastuzumab-EU would not be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less